CLINICAL TRIAL: NCT06189235
Title: Development of Ultrasonography-guided Real-time Intelligent Monitoring, Evaluation and Biofeedback Training Modular Systems for Hand Therapy
Brief Title: Ultrasonography-guided Real-time Modular Systems for Hand Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B-ER-111-012
Record Dates: First submitted 2023-06-23; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-06

CONDITIONS: Health Adults; Patients With Traumatic Hand Injury
Keywords: Ultrasonography-guided; Biofeedback; Hand therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- System development: Validation for patients (No Intervention): No intervention. The patients will receive one time of MRI and three times of ultrasound evaluation on the injured area, each evaluaitons will be done by two to three days interval.
- System development: Building dataset from healthy subjects (No Intervention): No intervention. The healthy subjects will receive one time of ultrasound evaluation on the dominant hand, the different part and different axis in dominant hand will be assessed in types of images or films for building the dataset.
- System application: Understanding the recovery patterns in patients (No Intervention): No intervention. The patients will receive three times of ultrasound evaluation on the injured area and hand function assessments, each evaluaitons will be done by two weeks interval.
- System application: Biofeedback training (Experimental): The program last for one month. In this program, the patients receive traditional rehabilitation protocol assigned from original hospital or therapist. Also, ultrasound evaluation and hand function assessment will be performed at pre-test, one follow-up test and post-test, which will be done with two weeks interval.
  For this biofeedback training group, the therapist and patients will be asked to use the hint recommanded by modular system to assist the rehabilitation excepting the traditional routine at least two times a week.
  Interventions: Other: Biofeedback training
- System application: Traditional training (No Intervention): The program last for one month. In this program, the patients receive traditional rehabilitation protocol assigned from original hospital or therapist. Also, ultrasound evaluation and hand function assessment will be performed at pre-test, one follow-up test and post-test, which will be done with two weeks interval.

INTERVENTIONS:
Other: Biofeedback training — The target of additional biofeedback training is to provide hints which are related to the essential aspects during hand therapy such as the stress on the tissue and the distance of tendon gliding.
  Arms: System application: Biofeedback training

SUMMARY:
This study aimed to develop an ultrasonography-guided real-time modular system and try to apply it to clinical hand therapy using.

This study was divided into two parts. The first part is an observational study design. The ultrasonography-guided real-time modular system will be developed and integrated, and its overall reliability and validity will be tested in this part. Once the software and hardware of the modular system has been established, numerous hand-related ultrasonography data will be collected for building an artificial intelligence model for detecting the anatomic structures in hand, evaluating the status of the tissues in hand.

The second part is an interventional study design. The clinical application of the modular system on hand injured patients is conducted, and the biofeedback mechanics will also be defined in the second part. The patients will be recruited into the research to receive both traditional rehabilitation and the one which combines with biofeedback training via the modular system. The effect of the traditional and biofeedback-added rehabilitation will be compared.

ELIGIBILITY:
【Patients】

Inclusion Criteria:

* Traumatic hand injury (distal from wrist joint above 8 weeks and within one year)
* Able to do active motion and resistive activities
* Understand and cooperate the experiment

Exclusion Criteria:

* Burn, amputees or has history of arthritis
* Combined with other central or peripheral nerve deficits which cause difficulty in movements

【Healthy subjects】

Inclusion Criteria:

* No history of traumatic hand injury and other hand related conditions
* Understand and cooperate the experiment

Exclusion Criteria:

* Burn, amputees or has history of arthritis
* Combined with other central or peripheral nerve deficits which cause difficulty in movements

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 149 (Estimated)
Dates: Start 2023-06-28 (Actual); Primary Completion 2024-04-26 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in tissue characteristics - Ultrasonography platform - Hand Injuries Group (System development) - Baseline | Baseline, 2-3 days after baseline, 4-5 days after baseline
  An ultrasonography platform and different installed modes will be used to gather the images from affected and unaffected hand of patients with hand injuries. These data will be collected three times in hand injuries group to know how will the tissue change between different time points.
Change from Baseline tissue characteristics at 2-3 days - Ultrasonography platform - Hand Injuries Group (System development) - 2-3 days after baseline | Baseline, 2-3 days after baseline, 4-5 days after baseline
  An ultrasonography platform and different installed modes will be used to gather the images from affected and unaffected hand of patients with hand injuries. These data will be collected three times in hand injuries group to know how will the tissue change between different time points.
Change from Baseline tissue characteristics at 4-5 days - Ultrasonography platform - Hand Injuries Group (System development) - 4-5 days after baseline | Baseline, 2-3 days after baseline, 4-5 days after baseline
  An ultrasonography platform and different installed modes will be used to gather the images from affected and unaffected hand of patients with hand injuries. These data will be collected three times in hand injuries group to know how will the tissue change between different time points.
Ultrasonography platform - Healthy Group - Baseline | Baseline
  An ultrasonography platform and different installed modes will be used to gather the images and films from dominant hand of healthy adults for building the dataset.
Change in tissue characteristics - Ultrasonography platform - Hand Injuries Group (System application) - Baseline | Baseline, 2 weeks after baseline, 4 weeks after baseline
  An ultrasonography platform and different installed modes will be used to gather the images from affected and unaffected hand of patients with hand injuries. These data will be collected three times in hand injuries group to know how will the tissue change between different time points.
Change from Baseline tissue characteristics at 2 weeks - Ultrasonography platform - Hand Injuries Group (System application) - 2 weeks after baseline | Baseline, 2 weeks after baseline, 4 weeks after baseline
  An ultrasonography platform and different installed modes will be used to gather the images from affected and unaffected hand of patients with hand injuries. These data will be collected three times in hand injuries group to know how will the tissue change between different time points.
Change from Baseline tissue characteristics at 4 weeks - Ultrasonography platform - Hand Injuries Group (System application) - 4 weeks after baseline | Baseline, 2 weeks after baseline, 4 weeks after baseline
  An ultrasonography platform and different installed modes will be used to gather the images from affected and unaffected hand of patients with hand injuries. These data will be collected three times in hand injuries group to know how will the tissue change between different time points.
Change in joint ROM - Goniometer - Hand Injuries Group (System application) - Baseline | Baseline, 2 weeks after baseline, 4 weeks after baseline
  The goniometer will be used to measure the range of motion (ROM) in the affected and affected finger.
Change from Baseline joint ROM at 2 weeks - Goniometer - Hand Injuries Group (System application) - 2 weeks after baseline | Baseline, 2 weeks after baseline, 4 weeks after baseline
  The goniometer will be used to measure the range of motion (ROM) in the affected and affected finger.
Change from Baseline joint ROM at 4 weeks - Goniometer - Hand Injuries Group (System application) - 4 weeks after baseline | Baseline, 2 weeks after baseline, 4 weeks after baseline
  The goniometer will be used to measure the range of motion (ROM) in the affected and affected finger.
Change in single digit force - Force sensors - Hand Injuries Group (System application) - Baseline | Baseline, 2 weeks after baseline, 4 weeks after baseline
  A force sensor will be used to collect the single digit force data in affected and unaffected finger.
Change from Baseline single digit force at 2 weeks - Force sensors - Hand Injuries Group (System application) - 2 weeks after baseline | Baseline, 2 weeks after baseline, 4 weeks after baseline
  A force sensor will be used to collect the single digit force data in affected and unaffected finger.
Change from Baseline single digit force at 4 weeks - Force sensors - Hand Injuries Group (System application) - 4 weeks after baseline | Baseline, 2 weeks after baseline, 4 weeks after baseline
  A force sensor will be used to collect the single digit force data in affected and unaffected finger.
Change in grip and pinch force - Hand dynamometer - Hand Injuries Group (System application) - Baseline | Baseline, 2 weeks after baseline, 4 weeks after baseline
  Hand dynamometer will be used to measure the grip strength and pinch strength.
Change from Baseline grip and pinch force at 2 weeks - Hand dynamometer - Hand Injuries Group (System application) - 2 weeks after baseline | Baseline, 2 weeks after baseline, 4 weeks after baseline
  Hand dynamometer will be used to measure the grip strength and pinch strength.
Change from Baseline grip and pinch force at 4 weeks - Hand dynamometer - Hand Injuries Group (System application) - 4 weeks after baseline | Baseline, 2 weeks after baseline, 4 weeks after baseline
  Hand dynamometer will be used to measure the grip strength and pinch strength.
Change in hand dexterity - Purdue pegboard test - Hand Injuries Group (System application) - Baseline | Baseline, 2 weeks after baseline, 4 weeks after baseline
  The Purdue pegboard test will be used to test the unimanual and bimanual manipulation versus hand dexterity.
Change from Baseline hand dexterity at 2 weeks - Purdue pegboard test - Hand Injuries Group (System application) - 2 weeks after baseline | Baseline, 2 weeks after baseline, 4 weeks after baseline
  The Purdue pegboard test will be used to test the unimanual and bimanual manipulation versus hand dexterity.
Change from Baseline hand dexterity at 4 weeks - Purdue pegboard test - Hand Injuries Group (System application) - 4 weeks after baseline | Baseline, 2 weeks after baseline, 4 weeks after baseline
  The Purdue pegboard test will be used to test the unimanual and bimanual manipulation versus hand dexterity.
Change in perspective hand function - Disabilities of the Arm, Shoulder and Hand - Hand Injuries Group (System application) - Baseline | Baseline, 2 weeks after baseline, 4 weeks after baseline
  The Disabilities of the Arm, Shoulder and Hand (DASH) is a questionnaire, which will be used to evaluate disorders and measure disability of the upper extremities and monitor change or function over time.
Change from Baseline perspective hand function at 2 weeks - Disabilities of the Arm, Shoulder and Hand - Hand Injuries Group (System application) - 2 weeks after baseline | Baseline, 2 weeks after baseline, 4 weeks after baseline
  The Disabilities of the Arm, Shoulder and Hand (DASH) is a questionnaire, which will be used to evaluate disorders and measure disability of the upper extremities and monitor change or function over time.
Change from Baseline perspective hand function at 4 weeks - Disabilities of the Arm, Shoulder and Hand - Hand Injuries Group (System application) - 4 weeks after baseline | Baseline, 2 weeks after baseline, 4 weeks after baseline
  The Disabilities of the Arm, Shoulder and Hand (DASH) is a questionnaire, which will be used to evaluate disorders and measure disability of the upper extremities and monitor change or function over time.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng-Kung University Hospital, Tainan, Taiwan